CLINICAL TRIAL: NCT04043481
Title: Relation of the Peripheral Perfusion Index Derived From Pulse Oximetry to Modified Allen's Test in Evaluation of Hand Perfusion
Brief Title: Modified Allen's Test and Peripheral Perfusion Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Mostafa Esmaeil Osman, Principal Investigator, Assiut University
Other Study IDs: Perfusion index & Allen's test
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Perfusion
Keywords: Perfusion index; modified Allen's test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to detect the relation between results of the peripheral perfusion index and modified Allen's test.

DETAILED DESCRIPTION:
The modified Allen's test (MAT) is commonly used to assess hand perfusion. Other non-invasive methods including plethysmography, pulse oximetry and duplex ultrasonography are used nowadays. The perfusion index is calculated as the ratio of the pulsatile blood flow to non- pulsatile blood flow in peripheral tissue.

In this study, we will try to detect the relation between results of the peripheral perfusion index and modified Allen's test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients or healthy volunteers

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Perfusion of the hand using the perfusion index | Preoperative
Perfusion of the hand using the modified Allen's test | Preoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt